CLINICAL TRIAL: NCT03425994
Title: Efficacy and Safety of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (Genvoya) as Maintenance Treatment of HIV-1/Hepatitis B Virus (HBV)-Coinfected Patients: an Observational Study
Brief Title: Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide as Maintenance Treatment for HIV/HBV-coinfection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); National Taiwan University Hospital, Yun-Lin Branch (Other); Far Eastern Memorial Hospital (Other); Taoyuan General Hospital (Other Government); Mackay Memorial Hospital (Other); Chung Shan Medical University (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Changhua Christian Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); E-DA Hospital (Other); Lotung Poh-Ai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201710056RIPB
Record Dates: First submitted 2018-01-11; First posted 2018-02-08 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Hepatitis B in HIV Patient; Kidney Injury; Bone Diseases
MeSH Terms: conditions — Bone Diseases | interventions — elvitegravir; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide: Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (Genvoya) tablet by mouth, once daily for 48 weeks
  Interventions: Drug: Elvitegravir/Cobicistat/Emtricitabine

INTERVENTIONS:
Drug: Elvitegravir/Cobicistat/Emtricitabine — Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide 150mg/150mg/200mg/10mg (Genvoya) film coated tablet
  Other Names: Genvoya

SUMMARY:
Tenofovir alafenamide (TAF), active against both HIV and HBV, demonstrates similar antiviral efficacy but improved renal and bone safety compared to tenofovir disoproxil fumarate (TDF) in HIV-1-infected patients. HIV-1-infected patients whose estimated glomerular filtration rate (eGFR) between 30-69 mL/min were shown to have minimal change in eGFR and improved proteinuria, albuminuria, and bone mineral density after switching to a single-tablet regimen containing Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (EVG/cob/FTC/TAF). For treatment of chronic HBV infection, a similar proportion of HBV-monoinfected patients who received TAF and those who received TDF achieved undetectable HBV DNA at 48 weeks of therapy. Although TAF is effective for HIV and HBV suppression, data on efficacy of TAF are limited among patients co-infected with both viruses. Currently, only one open-label, single-arm study had investigated the efﬁcacy and safety of TAF in HIV/HBV-coinfected patients. In this study, 72 HIV/HBV-coinfected patients switching to EVG/cob/FTC/TAF were enrolled, and 91.7% of them maintained or achieved virologic suppression for both HIV and HBV at 48 weeks of therapy. Seroconversion occurred in 2.9% of HBsAg-positive participants and in 3.3% of HBeAg-positive participants. Improvements in eGFR and declines in markers of bone turnover of the participants were observed. The limitations of the above study are the small sample size. Taiwan is a country hyperendemic for HBV infection, with 19.8% of HIV-positive patients who were born before the implementation of nationwide neonatal vaccination in 1986 had concurrent chronic HBV infection. To further the understanding of the difference between TAF- and TDF-containing combination antiretroviral therapy among HIV/HBV-coinfected patients, the investigators plan to conduct an observational study to evaluate the efficacy and safety of EVG/cob/FTC/TAF as maintenance treatment of HIV/HBV-coinfected patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 20 years
* Diagnosed with HIV and HBV-coinfection. HBV infection is defined as positive HBsAg for 6 months or longer before enrollment of the study
* Serum HBV DNA load <9 log10 IU/mL
* On Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) or TDF plus lamivudine (3TC) as backbone plus a 3rd agent for HIV infection for 6 months or longer
* Plasma HIV RNA load <50 copies/mL twice over the past 12 months
* No known resistance mutations to Integrase strand transfer inhibitors (InSTIs), and no previous history of HIV treatment failure under InSTIs-containing combination antiretroviral therapy (cART). HIV treatment failure is defined as a plasma HIV RNA load >400 copies/mL after 6 months of InSTIs-containing cART.
* No known resistance mutations to TDF, 3TC, or FTC, and no previous history of HIV treatment failure while on TDF, 3TC, or FTC-containing cART. HIV treatment failure is defined as a plasma HIV RNA load >400 copies/mL after 6 months of TDF, 3TC, or FTC-containing cART.
* Baseline eGFR (estimated glomerular filtration rate) ≥30 mL/min per 1.73m2 (calculated by CKD-EPI equation)
* AST and ALT ≤2-fold the upper limit of normal
* Able to sign the written informed consent

Exclusion Criteria:

* Active opportunistic illness
* On treatment of tuberculosis
* Pregnancy or lactation
* Hepatic decompensation (Child-Pugh C)
* Allergic to TDF, TAF, 3TC, FTC, or InSTIs
* Intolerance of InSTIs
* Hepatitis C virus (HCV)-coinfection and plan to start treatment with direct-acting antiviral agents or interferon/ribavirin within 48 weeks
* Concurrent use of rifamycins, phenytoin, and other drugs that are contraindicated with EVG/cob/FTC/TAF

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/HBV-coinfected patients
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with undetectable plasma HBV DNA load | 48 weeks
  Proportion of patients achieving undetectable plasma HBV DNA load (defined as <128 copies/mL)

SECONDARY OUTCOMES:
Decreases of plasma HBV DNA load | 48 weeks
  Decreases of plasma HBV DNA load (in log10 copies/mL)
Proportion of patients with plasma HIV RNA load <50 copies/mL | 48 weeks
  Proportion of patients achieving plasma HIV RNA load <50 copies/mL
Liver function | 48 weeks
  Change of serum aspartate aminotransferase (AST) and alanine transaminase (ALT)
Number of patients with change of HBV serology markers | 48 weeks
  Number of patients with HBsAg loss, hepatitis B e-antigen (HBeAg) loss, or appearance of anti-HBs and anti-HBe
Serum creatinine | 48 weeks
  Changes of serum creatinine from baseline
Number of patients with an increase of serum creatinine | 48 weeks
  Number of patients with an increase of serum creatinine by ≥0.3 mg/dL or ≥50% from baseline
Estimated glomerular filtration rate | 48 weeks
  Changes of serum estimated glomerular filtration rate (eGFR, [mL/min per 1.73m2], calculated by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) from baseline
Number of patients with a decline of estimated glomerular filtration rate | 48 weeks
  Number of patients with a decline of estimated glomerular filtration rate (eGFR, calculated by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) by 15 mL/min per 1.73m2 or 20% from baseline
Urine protein-creatinine ratio | 48 weeks
  Change of urine protein-creatinine ratio (UPCR) from baseline
Urine albumin-creatinine ratio | 48 weeks
  Change of urine albumin-creatinine ratio (UACR) from baseline
Urine β-2 microglobulin | 48 weeks
  Change of β-2 microglobulin from baseline
Bone disease | 48 weeks
  Change of bone mineral density
Adverse drug reaction | 48 weeks
  Number and types of adverse drug reaction related to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sax PE, Wohl D, Yin MT, Post F, DeJesus E, Saag M, Pozniak A, Thompson M, Podzamczer D, Molina JM, Oka S, Koenig E, Trottier B, Andrade-Villanueva J, Crofoot G, Custodio JM, Plummer A, Zhong L, Cao H, Martin H, Callebaut C, Cheng AK, Fordyce MW, McCallister S; GS-US-292-0104/0111 Study Team. Tenofovir alafenamide versus tenofovir disoproxil fumarate, coformulated with elvitegravir, cobicistat, and emtricitabine, for initial treatment of HIV-1 infection: two randomised, double-blind, phase 3, non-inferiority trials. Lancet. 2015 Jun 27;385(9987):2606-15. doi: 10.1016/S0140-6736(15)60616-X. Epub 2015 Apr 15. PMID 25890673
- [Background] Pozniak A, Arribas JR, Gathe J, Gupta SK, Post FA, Bloch M, Avihingsanon A, Crofoot G, Benson P, Lichtenstein K, Ramgopal M, Chetchotisakd P, Custodio JM, Abram ME, Wei X, Cheng A, McCallister S, SenGupta D, Fordyce MW; GS-US-292-0112 Study Team. Switching to Tenofovir Alafenamide, Coformulated With Elvitegravir, Cobicistat, and Emtricitabine, in HIV-Infected Patients With Renal Impairment: 48-Week Results From a Single-Arm, Multicenter, Open-Label Phase 3 Study. J Acquir Immune Defic Syndr. 2016 Apr 15;71(5):530-7. doi: 10.1097/QAI.0000000000000908. PMID 26627107
- [Background] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Background] Gallant J, Brunetta J, Crofoot G, Benson P, Mills A, Brinson C, Oka S, Cheng A, Garner W, Fordyce M, Das M, McCallister S; GS-US-292-1249 Study Investigators. Brief Report: Efficacy and Safety of Switching to a Single-Tablet Regimen of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide in HIV-1/Hepatitis B-Coinfected Adults. J Acquir Immune Defic Syndr. 2016 Nov 1;73(3):294-298. doi: 10.1097/QAI.0000000000001069. PMID 27171740
- [Derived] Huang YS, Cheng CY, Liou BH, Lu PL, Cheng SH, Lee YT, Liu CE, Sun HY, Yang CJ, Tang HJ, Lin SP, Ho MW, Huang SH, Tsai HC, Lee CH, Hung CC; Taiwan HIV Study Group. Efficacy and Safety of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide as Maintenance Treatment in HIV/HBV-Coinfected Patients. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):473-481. doi: 10.1097/QAI.0000000000002589. PMID 33273214